CLINICAL TRIAL: NCT00897936
Title: A Pilot Study to Characterize the Genomic and Epigenomic Signature of NPM Positive Vs. NPM Negative NCL
Brief Title: DNA Analysis of Tumor Tissue From Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000476571; ECOG-E1900T2
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia in remission; recurrent adult acute myeloid leukemia; untreated adult acute myeloid leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22)
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Congenital Abnormalities | interventions — DNA Methylation; Comparative Genomic Hybridization; In Situ Hybridization, Fluorescence; Microarray Analysis; Polymerase Chain Reaction; Immunologic Techniques

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: DNA methylation analysis
Genetic: comparative genomic hybridization
Genetic: fluorescence in situ hybridization
Genetic: microarray analysis
Genetic: polymerase chain reaction
Other: diagnostic laboratory biomarker analysis
Other: immunologic technique

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how well patients respond to treatment.

PURPOSE: This laboratory study is looking at tissue samples from patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine gene expression, genome integrity, cytosine methylation, and chromatin structure in patients with normal cytogenetics leukemia (NCL) acute myeloid leukemia.
* Determine whether NCL can be deconstructed into specific disease entities by analysis of the integrated genomic and epigenomic datasets using supervised and unsupervised methods in these patients.
* Identify the gene pathways that define NCL subtypes and molecular targets for validation in preclinical and clinical trials for these patients.
* Determine whether integrated analysis provides markers of prognostic and therapeutic response that accurately predicts clinical outcome and can be used to select patients for risk-stratified therapeutic trials.

OUTLINE: This is a pilot, multicenter study.

Samples are analyzed to assess array comparative genomic hybridization using polymerase chain reaction (PCR) and fluorescent in situ hybridization; chromatin immunoprecipitations (chip) using PCR; Hpa II tiny fragment enrichment by ligation-mediated PCR (HELP) using DNA methylation analysis; and gene expression profiling.

PROJECTED ACCRUAL: A total of 32 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia
* Enrolled on clinical trial ECOG-E1900

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2006-03-23 (Actual); Primary Completion 2009-10-15 (Actual); Study Completion 2009-10-15 (Actual)

PRIMARY OUTCOMES:
Nucleophosmin exon 12 mutation-related normal cytogenetics leukemia (NCL) has a specific genetic and epigenetic profile | 1 day
Relatedness on a per-gene basis of cross-platform data | 1 day
Ability of supervised clustering to distinguish subgroups according to clinical prognostic and biomarker indicators | 1 day
Ability of unsupervised clustering to identify subgroups of NCL patients | 1 day
Relative power of each platform mentioned above vs the integrated platforms | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Ari M. Melnick, MD, Study Chair — Albert Einstein College of Medicine